CLINICAL TRIAL: NCT00882232
Title: Transperineal Injection of Cross-linked Hyaluronan Gel Into Anterior Perirectal Fat to Reduce Rectal Toxicity From High Dose Rate Brachytherapy and/or Intensity-Modulated Radiation Therapy for Prostate Cancer
Brief Title: Cross-linked Hyaluronan Gel Reduces Rectal Toxicity Due to Radiation Therapy for Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Center of Irvine (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G080064; S002
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer; cross-linked; hyaluronan; gel; Hylaform; rectal; toxicity
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Cross-linked hyaluronan gel and radiotherapy. Cross-linked hyaluronan gel is injected under anesthesia between the prostate and rectum prior to the start of radiotherapy. The gel pushes the prostate away from the rectum over several months, thereby reducing the dose of radiation delivered to the rectum. Hyaluronic acid is a naturally-occurring substance that is gradually absorbed by the body.
  Interventions: Device: Cross-linked hyaluronan gel

INTERVENTIONS:
Device: Cross-linked hyaluronan gel — Single, transperitoneal injection of 9 mL cross-linked hyaluronan gel into anterior perirectal fat under anesthesia. The gel is injected prior to the start of radiotherapy and is absorbed by the body over several months. It increases the seapartion between the prostate and rectum by 1/3" to 2/3" at the start of radiotherapy.
  Other Names: Hylaform

SUMMARY:
The primary purpose of this study is to determine if cross-linked hyaluronan gel reduces the dose of radiation delivered to the rectum and the rectal toxicity of radiotherapy for localized prostate cancer.

DETAILED DESCRIPTION:
The main risk associated with transperineal injection of cross-linked hyaluronan gel into the anterior perirectal fat is infection. Prophylactic antibiotics will be given, resulting in a <5% risk. Another possible risk (<5%) is an allergic reaction such as itching. Patients who are allergic to avian products will be excluded from the study. Tenderness and pain at the injection site are possible. Bleeding, bruising, redness, or discoloration or the formation of a bump (granuloma) or scar (keloid) at the injection site is also possible. Embolization of cross-linked hyaluronan gel through the blood is a potential, rare complication if the gel is injected into a blood vessel rather than into fat. Prada et al. did not see any side effects related to the injection or the material itself in 27 patients based on a mean follow-up of 13 months (range: 9-22 months). Patients did not complain of pain, tenesmus, rectal pressure, or a sensation of rectal filling. Risks beyond 22 months are not well defined. Potential benefits of cross-linked hyaluronan gel include fewer rectal complications due to radiotherapy for early-stage prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed adenocarcinoma of the prostate, clinical stage T1c-T2c, NX, N0, M0.
2. Nodes determined to be negative by imaging methods will be classified as NX. Only nodes determined to be negative by surgical sampling will be classified as N0.
3. Prostate cancer biopsy grading by Gleason score classification is mandatory.
4. No prior pelvic radiotherapy. Induction hormonal therapy for less than or equal to 6 months is acceptable.
5. Prostate volume by TRUS < 50 cc prior to HDR brachytherapy.
6. Prostate specific antigen (PSA) less than or equal to 30 ng/ml.
7. Patient has provided informed consent.

Exclusion Criteria:

1. Clinical stage T3 or T4.
2. Clinical evidence of lymph node involvement (N1).
3. Clinical evidence of distant metastases (M1).
4. Radical surgery for carcinoma of the prostate.
5. Allergy to avian products.
6. Significant mental, medical, or physical impairment.
7. Prisoners.
8. Employees of the Cancer Center of Irvine.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Mean rectal dose without Hylaform vs with Hylaform | 8 months

SECONDARY OUTCOMES:
Severity of late diarrhea without Hylaform vs with Hylaform | 33 months
Rectal wall relative V60 and V70 without Hylaform vs with Hylaform | 8 months
Severity of acute diarrhea during IMRT without Hylaform vs with Hylaform | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Tokita, MD, Principal Investigator — Cancer Center of Irvine; Richard B Wilder, MD, Study Director — Cancer Center of Irvine
Locations (1):
- Cancer Center of Irvine, Irvine, California, United States